CLINICAL TRIAL: NCT05119972
Title: A Multi-center, Phase Ib/IIa Clinical Trial to Evaluate the Tolerability, PK and Efficacy of ZSP1603 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Tolerability, Pharmacokinetics and Efficacy of ZSP1603 in Patients With Idiopathic Pulmonary Fibrosis （IPF）
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZSP1603-20-02
Record Dates: First submitted 2021-10-09; First posted 2021-11-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial has two parts, a part 1 and a part 2, in part 1 will be unblinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- part1:ZSP1603 dose1 (Experimental)
  Interventions: Drug: ZSP1603
- part1:ZSP1603 dose2 (Experimental)
  Interventions: Drug: ZSP1603
- part1:ZSP1603 dose3 (Experimental)
  Interventions: Drug: ZSP1603
- Part2: ZSP1603 dose (Experimental)
  Interventions: Drug: ZSP1603
- Part2: placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZSP1603 — ZSP1603 administered orally
  Arms: Part2: ZSP1603 dose; part1:ZSP1603 dose1; part1:ZSP1603 dose2; part1:ZSP1603 dose3
Drug: Placebo — Placebo administered orally
  Arms: Part2: placebo

SUMMARY:
This study was divided into two parts. The first part was a dose escalation study: a open label dose escalation design was used to evaluate the safety, tolerance and pharmacokinetic characteristics of ZSP1603 in IPF patients. The second part was a randomized double-blind placebo-controlled design was used to preliminatively investigate the efficacy and safety of ZSP1603 in the treatment of IPF at the target dose.

ELIGIBILITY:
Inclusion Criteria:

* IPF diagnosed, according to 2018 American Thoracic Society (ATS), European Respiratory Society (ERS), Japanese Respiratory Society (JRS), Latin American Thoracic Association (ALAT) IPF guideline for diagnosis and management;
* Dlco (corrected for Hb): 30%-79% predicted of normal;
* FVC>= 50% predicted of normal;

Exclusion Criteria:

* FEV1/FVC< 0.7;
* PaO2 in resting state without oxygen inhalation < 50mmHg;
* Subjects who were likely to be lung transplant recipients or expected to survive less than 1 year during the study period as assessed by the investigator;
* Poorly controlled cardiovascular and cerebrovascular diseases;
* Patients who had used nidanib, pirfenidone, interferon, n-acetylcysteine, azathioprine, cyclophosphamide, cyclosporine, prednisone > 15mg/ day (or equivalent dose of other glucocorticoids) within 4 weeks before enrollment; Those who had used Chinese herbal medicine or acupuncture treatment within 1 week before enrollment;

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to 16 weeks
  TEAEs will be summarized displaying the number of TEAEs along with the number and percentage of participants with at least one TEAE according to: Number of AEs, Severity and relation to study drug.
Plasma concentrations of ZSP1603 | up to 15 Days
  Pharmacokinetic analysis

SECONDARY OUTCOMES:
Change in FVC From Baseline at 12 weeks | up to 12 weeks
  Change of Forced Vital Capacity (FVC) evaluated from baseline until 12 weeks of treatment.
Change in FVC%Pred from baseline at 12 weeks | up to12 weeks
  Change of predicted Forced Vital Capacity (FVC) (% Predicted) evaluated from baseline until 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Lung Hospital, Shanghai, Shanghai Municipality, China